CLINICAL TRIAL: NCT03775850
Title: A Phase I Open-label Study of EDP1503 Alone and in Combination With Pembrolizumab in Patients With Advanced Metastatic Colorectal Carcinoma, Triple-negative Breast Cancer, and Checkpoint Inhibitor Relapsed Tumors
Brief Title: A Study of EDP1503 in Patients With Colorectal Cancer, Breast Cancer, and Checkpoint Inhibitor Relapsed Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDP1503-101; KEYNOTE-939 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer Metastatic; Triple Negative Breast Cancer; Non Small Cell Lung Cancer; Bladder Cancer; GastroEsophageal Cancer; Renal Cell Carcinoma; MSI-H
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of three cohorts based on disease condition: Cohort A (microsatellite stable colorectal cancer); Cohort B (Triple negative breast cancer); Cohort C (PD-1 relapsed tumors: non small cell lung cancer, gastroesophageal cancer, or any microsatellite unstable or renal cell carcinoma). Patients will receive monotherapy with EDP1503 for a period of 2 weeks, following which they will be dosed with a combination of EDP1503 and pembrolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Cohort A includes patients with microsatellite stable (MSS) colorectal cancer (CRC). Patients will receive a 14 day run-in of EDP1503 alone, following which they will be treated with a combination of EDP1503 and pembrolizumab.
  Interventions: Biological: EDP1503; Biological: Pembrolizumab
- Cohort B (Experimental): Cohort B includes patients with Triple Negative Breast Cancer (TNBC). Patients will receive a 14 day run-in of EDP1503 alone, following which they will be treated with a combination of EDP1503 and pembrolizumab.
  Interventions: Biological: EDP1503; Biological: Pembrolizumab
- Cohort C (Experimental): Cohort C includes patients with non-small-cell lung cancer (NSCLC), bladder cancer; gastroesophageal (GE) cancer, any microsatellite unstable, or renal cell carcinoma (RCC) who are relapsed to prior PD-1/L1 therapy. Patients will receive a 14 day run-in of EDP1503 alone, following which they will be treated with a combination of EDP1503 and pembrolizumab.
  Interventions: Biological: EDP1503; Biological: Pembrolizumab

INTERVENTIONS:
Biological: EDP1503 — 4 capsules taken by mouth twice daily. Each capsule will contain ≥ 7.5x10^10 colony-forming units (CFU)
Biological: Pembrolizumab — 200 mg given by intravenous (IV) infusion once every 3 weeks
  Other Names: Keytruda

SUMMARY:
This study is being conducted to assess the safety, tolerability, and efficacy of EDP1503 alone and in combination with pembrolizumab in patients with advanced metastatic colorectal carcinoma, triple-negative breast cancer, and checkpoint inhibitor relapsed tumors

DETAILED DESCRIPTION:
This will be a Phase I open-label study which will involve a 2-week monotherapy with EDP1503, following which the patients will be dosed with a combination of EDP1503 and pembrolizumab.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors who have had disease progression after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment.
2. Have adequate organ function as defined in the clinical protocol. Specimens must be collected within 10 days prior to the start of study treatment.
3. Have provided an archival tumor tissue sample obtained since the most recent prior anticancer regimen or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
4. Measurable disease by RECIST v1.1 as assessed by the local site investigator/radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Metastatic disease not suitable for upfront curative-intent surgery.
6. Progressive disease on previous line of therapy per treating investigator (additional specific criteria for cohort C).
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
8. Additional tumor-specific inclusion criteria

Selected Exclusion Criteria:

1. Has received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
2. Treatment with investigational therapy within 28 days prior to initiation of study treatment.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE).
4. Has received prior systemic anti-cancer therapy within 28 days or 5 half-lives, whichever is shorter prior to treatment.

   Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy may be eligible.

   Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
5. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   1. Unstable angina or acute myocardial infarction ≤ 3 months prior to C1D1;
   2. Clinically significant heart disease (e.g., symptomatic congestive heart failure [e.g., >NYHA Class 2]; uncontrolled arrhythmia, or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen).
6. Uncontrolled active severe systemic infection requiring parenteral antibiotics within 1 week, and systemic antivirals or antifungals within two weeks prior to C1D1.
7. Patients with active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
8. Patients with severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Prior malignancies:

   1. Patients with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (i.e. cervix, breast) may enroll irrespective of the time of diagnosis.
   2. Patients with a known additional malignancy that is progressing or has required active treatment within the past which may interfere with the interpretation of the study. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Sponsor. Cancer treated with curative intent > 5 years previously and without evidence of recurrence will be allowed.
10. Patients with a diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
11. Patients with uncontrolled vomiting or dirrahea that could interfere with the GI exposure to EDP1503.
12. Patients who are transfusion dependent should be discussed with the Medical Monitor
13. Patients unwilling to comply with the protocol including required biopsies and sample collections required to measure disease.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has received a live vaccine within 30 days of planned C1D1. Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed. Intranasal influenza vaccines (e.g FluMist) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of EDP1503 alone and in combination with pembrolizumab as assessed per CTCAE v5.0 | 2 years
  Number of participants with EPD1503 related adverse events as assessed per CTCAE v5.0
Safety and tolerability of EDP1503 alone and in combination with pembrolizumab | 2 years
  Safety and tolerability of EDP1503 alone and in combination with pembrolizumab assessed via clinical laboratory evaluations
Evidence of anti-tumor activity of EDP1503 based on ORR | 2 years
  To determine preliminary evidence of anti-tumor activity of EDP1503 in patients

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  Progression Free Survival
Overall Survival | 2 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (8):
- United States (5):
  - Highlands Oncology Group, Rogers, Arkansas
  - Florida Cancer Specialists, Sarasota, Florida
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
- Canada (3):
  - Centre de Recherche du CHUM, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang JS, Arrowsmith ER, Beck JT, Friedmann J, Jamal R, McHale D, Gardner H, Chisamore MJ, Ulahannan SV. Phase 1/2, open-label study of oral bacterial supplementation (EDP1503) plus pembrolizumab in participants with advanced or metastatic microsatellite-stable colorectal cancer, triple-negative breast cancer, and checkpoint inhibitor-relapsed tumors. Invest New Drugs. 2025 Aug;43(4):894-903. doi: 10.1007/s10637-025-01573-0. Epub 2025 Aug 20. PMID 40830709